CLINICAL TRIAL: NCT05700019
Title: Effects of 'Pinkwashed' Alcohol Ads in an Online RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-2338
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Standard Advertisements (Other): In the control condition, participants will view 3 advertisements for alcohol (shown in random order) that do not mention breast cancer awareness or charities. Advertisements will be real social media posts used by alcohol companies, modified only to remove dates, likes/comments, and references to specific geographic locations.
  Interventions: Behavioral: Control - Standard Advertisements
- Pinkwashed Advertisements (Experimental): In the pinkwashed condition, participants will view 3 advertisements for alcohol (shown in random order) that associate the alcohol company with breast cancer awareness or research (e.g., indicate that a portion of sales will be directed to a breast cancer-related foundation). Advertisements will be real social media posts used by alcohol companies, modified only to remove dates, likes/comments, and references to specific geographic locations.
  Interventions: Behavioral: Pinkwashed Advertisements

INTERVENTIONS:
Behavioral: Pinkwashed Advertisements — Real advertisements from alcoholic beverage companies' social media accounts that contain messaging or other features that associate the alcohol company with breast cancer awareness or research.
  Arms: Pinkwashed Advertisements
Behavioral: Control - Standard Advertisements — Real advertisements from the same alcoholic beverage companies' social media accounts that do not contain messaging or other features associated with breast cancer awareness or research.
  Arms: Control - Standard Advertisements

SUMMARY:
The primary objective of this study is to examine how exposure to "pinkwashed" alcohol advertisements (i.e., ads that associate the company with breast cancer awareness or charities) affects consumers' perceptions that alcohol increases the risk of breast cancer. The investigators will randomize participants to view 3 'pinkwashed' social media advertisements for alcohol or 3 control advertisements for alcohol (i.e., 'de-pinked' standard alcohol advertisements that match the intervention advertisements on overall design but do not mention breast cancer). Each participant will view the 3 advertisements for their arm (presented in random order) and respond to survey questions programmed in Qualtrics.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older

Exclusion Criteria:

* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Breast cancer risk perceptions | During ~20 minute online survey
  This outcome will be measured with an adapted item from the HINTS (2020) survey. The question is worded " In your opinion, how much does drinking [wine/beer/liquor] affect the risk of developing each of the following outcomes... Breast cancer." Response options are on a five point likert-type scale ranging from "Decreases risk a lot" (=1) to "Increases risk a lot " (=5). Participants will be asked to respond to this item three times, once for each type of alcoholic beverage presented (wine, beer, liquor). Scores from the three items will then be averaged for analyses. Higher scores indicate higher risk perceptions.

SECONDARY OUTCOMES:
Perceived product healthfulness | During ~20 minute online survey
  This outcome will be measured with one item adapted from Bollard et al (2016). The question will read: "How healthy or unhealthy do you think it is to drink this product?" and will be measured with a 5-point likert-type response scale ranging from "Very unhealthy" (1) to "Very healthy"(5). Higher scores indicate greater healthfulness perceptions.
Perceived social responsibility of brand | During ~20 minute online survey
  This outcome will be measured with one item adapted from Nan & Heo (2017). The question will read: "How socially responsible do you think the company that makes this product is?" and will be measured with a 5-point likert-type response scale ranging from "Very socially irresponsible" (1) to "Very socially responsible" (5). Higher scores indicate perceptions of social responsibility.
Favorable attitudes toward brand | During ~20 minute online survey
  This outcome will be measured with one item adapted from Nan & Heo (2017). The question will read: "How do you feel about the company that makes this product?" and will be measured with a 5-point likert-type response scale ranging from "Dislike it a lot" (1) to "Like it a lot" (5). Higher scores indicate more favorable attitudes.
Purchase intentions | During ~20 minute online survey
  This outcome will be measured with one item adapted from Hall et al (2020). The question will display all three advertisements that the participant was exposed to (either pinkwashed or control). It will then query: "How likely would you be to buy any of these products in the next 4 weeks, if they were available?" and will be measured with a 5-point likert-type response scale ranging from "Not at all likely" (1) to "Extremely likely" (5). Higher scores indicate greater purchase intentions.
Perceived misleadingness of ads | During ~20 minute online survey
  Measure of how misleading a participant perceives the advertisement. Assessed with 1 item adapted from Hall et al. 2020
Support for breast cancer warnings | During ~20 minute online survey
  Measure of participant support of including breast cancer warning labels on alcoholic beverage products. Assessed with 1 item adapted from Hall et al. 2018
Stomach cancer risk perceptions | During ~20 minute online survey
  This outcome will be measured with an adapted item from the HINTS (2020) survey. The question is worded " In your opinion, how much does drinking [wine/beer/liquor] affect the risk of developing each of the following outcomes... Stomach cancer." Response options are on a five point likert-type scale ranging from "Decreases risk a lot" (=1) to "Increases risk a lot " (=5). Participants will be asked to respond to this item three times, once for each type of alcoholic beverage presented (wine, beer, liquor). Scores from the three items will then be averaged for analyses. Higher scores indicate higher risk perceptions.
Mouth and throat cancer risk perceptions | During ~20 minute online survey
  This outcome will be measured with an adapted item from the HINTS (2020) survey. The question is worded " In your opinion, how much does drinking [wine/beer/liquor] affect the risk of developing each of the following outcomes... Mouth and throat cancer." Response options are on a five point likert-type scale ranging from "Decreases risk a lot" (=1) to "Increases risk a lot " (=5). Participants will be asked to respond to this item three times, once for each type of alcoholic beverage presented (wine, beer, liquor). Scores from the three items will then be averaged for analyses. Higher scores indicate higher risk perceptions.
Liver cancer risk perceptions | During ~20 minute online survey
  This outcome will be measured with an adapted item from the HINTS (2020) survey. The question is worded " In your opinion, how much does drinking [wine/beer/liquor] affect the risk of developing each of the following outcomes... Liver cancer." Response options are on a five point likert-type scale ranging from "Decreases risk a lot" (=1) to "Increases risk a lot " (=5). Participants will be asked to respond to this item three times, once for each type of alcoholic beverage presented (wine, beer, liquor). Scores from the three items will then be averaged for analyses. Higher scores indicate higher risk perceptions.
Liver disease risk perceptions | During ~20 minute online survey
  This outcome will be measured with an adapted item from the HINTS (2020) survey. The question is worded " In your opinion, how much does drinking [wine/beer/liquor] affect the risk of developing each of the following outcomes... Liver disease." Response options are on a five point likert-type scale ranging from "Decreases risk a lot" (=1) to "Increases risk a lot " (=5). Participants will be asked to respond to this item three times, once for each type of alcoholic beverage presented (wine, beer, liquor). Scores from the three items will then be averaged for analyses. Higher scores indicate higher risk perceptions.
Hypertension risk perceptions | During ~20 minute online survey
  This outcome will be measured with an adapted item from the HINTS (2020) survey. The question is worded " In your opinion, how much does drinking [wine/beer/liquor] affect the risk of developing each of the following outcomes...Hypertension." Response options are on a five point likert-type scale ranging from "Decreases risk a lot" (=1) to "Increases risk a lot " (=5). Participants will be asked to respond to this item three times, once for each type of alcoholic beverage presented (wine, beer, liquor). Scores from the three items will then be averaged for analyses. Higher scores indicate higher risk perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Marissa G Hall, PhD, Principal Investigator — UNC-Chapel Hill; Anna H Grummon, PhD, Principal Investigator — Stanford Univeristy; Kurt Ribsl, PhD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- UNC - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share our deidentified individual participant data, as well as our statistical analysis plan and analytic code on Open Science Framework (OSF), a publicly available data repository.
Supporting Information: SAP, Analytic Code
Time Frame: The deidentified dataset, SAP, and analytic code will be posted to OSF within 6 months of results publication. Materials will be available for 7 years after initial posting.
Access Criteria: There will be no access criteria; information will posted on a publicly available repository.
URL: http://osf.io/

REFERENCES:
- [Background] Nan X, Heo K. Consumer Responses to Corporate Social Responsibility (CSR) Initiatives: Examining the Role of Brand-Cause Fit in Cause-Related Marketing. Journal of Advertising. 2007;36(2):63-74. doi:10.2753/JOA0091-3367360204
- [Background] Hall MG, Lazard AJ, Grummon AH, Mendel JR, Taillie LS. The impact of front-of-package claims, fruit images, and health warnings on consumers' perceptions of sugar-sweetened fruit drinks: Three randomized experiments. Prev Med. 2020 Mar;132:105998. doi: 10.1016/j.ypmed.2020.105998. Epub 2020 Jan 23. PMID 31982477
- [Background] Bollard T, Maubach N, Walker N, Ni Mhurchu C. Effects of plain packaging, warning labels, and taxes on young people's predicted sugar-sweetened beverage preferences: an experimental study. Int J Behav Nutr Phys Act. 2016 Sep 1;13(1):95. doi: 10.1186/s12966-016-0421-7. PMID 27580589
- [Background] Hall MG, Marteau TM, Sunstein CR, Ribisl KM, Noar SM, Orlan EN, Brewer NT. Public support for pictorial warnings on cigarette packs: an experimental study of US smokers. J Behav Med. 2018 Jun;41(3):398-405. doi: 10.1007/s10865-018-9910-2. Epub 2018 Feb 6. PMID 29411272
- See also: HINTS survey items — https://hints.cancer.gov/